CLINICAL TRIAL: NCT06467630
Title: Prospective, National, Multicentre and Observational Clinical Investigation of R.T.R.+ Membrane Used in Guided Tissue Regeneration (GTR) in Dental Surgical Procedures
Brief Title: Measurement of the Performance and Safety of RTR+Membrane in Guided Tissue Regeneration (GTR) in Dental Surgical Procedures
Acronym: ObsR+
Status: Recruiting | Type: Observational
Sponsor: Septodont (Industry)
Responsible Party: Sponsor
Other Study IDs: RTR+ 2023-01
Record Dates: First submitted 2024-01-02; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-05

CONDITIONS: Guided Bone Regeneration
Keywords: Guided Bone Regeneration; Dental surgical procedures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Post-extraction socket preservation group: The 30 eligible patients are any male and female, adult patients with the following dental treatment to be done with the study device: Post-extraction socket preservation (not done concomitantly to implant placement).
  Interventions: Procedure: Preserving alveolar bone volume after tooth extraction
- Alveolar ridge augmentation group: The 30 eligible patients are any male and female, adult patients with the following dental treatment to be done with the study device: Alveolar ridge augmentation (not done concomitantly to implant placement).
  Interventions: Procedure: Alveolar crest reconstruction
- Guided Tissue Regeneration (GTR) during immediate implant placement group: The 30 eligible patients are any male and female, adult patients with the following dental treatment to be done with the study device: Guided Tissue Regeneration (GTR) during immediate implant placement
  Interventions: Procedure: Covering bone defects during immediate implant placement.

INTERVENTIONS:
Procedure: Preserving alveolar bone volume after tooth extraction — * Visit 1: A periodontal or dental implant surgery is done aiming to preserve alveolar bone volume after extraction
  * Visit 2 (10 days ± 4 days) - Early post-surgery follow-up
  * V2bis (1 month +/- 1 week) - Early post-surgery follow-up
  * Visit 3 (5 months ± 1 month) - Late post-surgery follow-up
  Groups: Post-extraction socket preservation group
Procedure: Alveolar crest reconstruction — * Visit 1: A periodontal or dental implant surgery is done aiming to alveolar crest reconstruction
  * Visit 2 (10 days ± 4 days) - Early post-surgery follow-up
  * Visit 3 (5 months ± 1 month) - Late post-surgery follow-up
  Groups: Alveolar ridge augmentation group
Procedure: Covering bone defects during immediate implant placement. — * Visit 1: A periodontal or dental implant surgery is done aiming to cover bone defects during immediate implant placement.
  * Visit 2 (10 days ± 4 days) - Early post-surgery follow-up
  * Visit 3 (3 months ± 1 month) - Late post-surgery follow-up
  Groups: Guided Tissue Regeneration (GTR) during immediate implant placement group

SUMMARY:
The goal of this observational study is to measure in real practice the performance and safety of RTR+Membrane, a synthetic dental membrane for guided tissue regeneration in periodontal or dental implant surgery. The main question it aims to answer is to measure the post-operative wound healing several months after surgery. Participants will be followed after their dental surgery via clinical examination and radiological and photos images.

DETAILED DESCRIPTION:
Participants are any adult patients with one of the 3 following dental treatments to be done with RTR+Membrane:

* post-extraction socket preservation,
* alveolar ridge augmentation,
* Guided Tissue Regeneration (GTR) during immediate implant placement.

Since it is a real-life evidence study in current practice, patients will be followed at their surgery and their follow-ups. Below are listed visits and type of data collected.

* V1 - Surgery: Demography, Medical history and concomitant treatments, Clinical/technical information (tooth extraction, surgery, membrane and grafting materials use), Clinical Exam, Photography, X-rays or Cone Beam Computed Tomography (CBCT)
* V2 - Early follow-up (including suture removal, if needed): Clinical Exam, Questionnaire, Photography
* V2bis - Early follow-up: Clinical Exam, Photography
* V3 - Late follow-up: Clinical Exam, Photography, X-rays or CBCT, Questionnaire

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult patient
* Patient with one of the 3 following dental treatments to be done with the study device: post-extraction socket preservation, alveolar ridge augmentation, or Guided Tissue Regeneration (GTR) during immediate implant placement.
* Patient affiliated or beneficiary of a social security system.
* Patient has signed his/her informed consent form.

Exclusion Criteria:

* Pregnancy or lactation
* Active tissue infection at the implant site
* Several dental treatments done simultaneously in non-contiguous dental zones
* Heavy smoker (>10 cigarettes / day)
* Patient receiving long-term corticosteroid therapy, anti-rejection drugs, bisphosphonates, head & neck radiotherapy or chemotherapy
* Patient with chronic infections (such as osteomyelitis) at the surgical site
* Patient with poorly controlled metabolic disorders (such as diabetes, osteomalacia, thyroid disorders)
* Patient with an auto-immune disease
* Patient under tutelage, vulnerable person, person without liberty, or unable to complete questionnaire independently

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are any male and female, adult patients with one of the 3 following dental treatments to be done with the study device:
  * post-extraction socket preservation*,
  * alveolar ridge augmentation*,
  * Guided Tissue Regeneration (GTR) during immediate implant placement.
  The dental treatment under investigation for one patient could be related to:
  * 1 alveolar socket corresponding to only 1 tooth;
  * 1 implant to be placed in replacement of 1 tooth;
  * several contiguous alveolar sockets;
  * Or, several contiguous implants to be placed. Dental treatments done simultaneously in non-contiguous dental zones won't be considered for this study.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-02-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Post-operative wound healing measured by the Early Wound-Healing Index | up to 6 months
  For all groups
  The Early Wound-Healing Index (EHI) has the following best to worst scoring:
  (EHI) 1: complete flap closure without fibrin line in the interproximal area. (EHI) 2: complete flap closure with fine fibrin line in the interproximal area. (EHI) 3: complete flap closure with fibrin clot in the interproximal area. (EHI) 4: incomplete flap closure with partial necrosis of the interproximal tissue. (EHI) 5: incomplete flap closure with complete necrosis of the interproximal tissue.
  The EHI is evaluated at the Visit 3 (late post-surgery follow-up) for the primary outcome measure.

SECONDARY OUTCOMES:
Post-operative wound healing measured by Early Wound-Healing Index | up to 14 days
  For all groups
  The Early Wound-Healing Index (EHI) has the following best to worst scoring:
  (EHI) 1: complete flap closure without fibrin line in the interproximal area. (EHI) 2: complete flap closure with fine fibrin line in the interproximal area. (EHI) 3: complete flap closure with fibrin clot in the interproximal area. (EHI) 4: incomplete flap closure with partial necrosis of the interproximal tissue. (EHI) 5: incomplete flap closure with complete necrosis of the interproximal tissue.
  The EHI is evaluated at the Visit 2 for this secondary outcome measure.
Post-operative wound healing measured by Early Wound Healing Score | up to 14 days
  For all groups
  The Early Wound Healing Score is from 0 (worse) to 10 (best).
  The EHS is evaluated at the Visit 2 for this secondary outcome measure.
Post-operative clinical exam | up to 6 months
  For all groups
  This is a descriptive secondary outcome measured by the investigator via the reporting of the presence or the absence of:
  * pain,
  * discomfort,
  * inflammation,
  * hematoma, redness,
  * swelling/suppuration,
  * membrane exposure,
  * dehiscence.
  The evaluation is done at visit 2, visit 2Bis, and visit 3.
Number of adverse device effects (at least possibly) related to study device | up to 6 months
  For all groups
Oral Health-Related Quality of Life measured by the Oral Health Impact Profile (OHIP-5 items) | up to 6 months
  For all groups
  The 5 items of OHIP are: Difficulty chewing any foods; Painful aching in the mouth; Felt uncomfortable about the appearance of teeth; Less flavor in the food; and, Difficulty doing the usual jobs.
  Score is from 0 (best) to 20 (worse). The evaluation is done at visit 2 and visit 3.
Radiological measurements on CBCT | up to 6 months
  Only for Post-extraction socket preservation sub-group & for Alveolar ridge augmentation sub-group
  The treatment efficacy is measured via the following measures on CBCT:
  A. Osseous changes in mesiodistal width of the alveolar ridge
  B. Osseous changes in height of the alveolar ridge
  C. Osseous changes in vestibulolingual dimension of the alveolar ridge.
  These changes are evaluated from Baseline to Visit 3.
Radiological measurements on retro-alveolar radios | up to 4 months
  Only for Guided Tissue Regeneration (GTR) during immediate implant placement subgroup.
  The treatment efficacy is measured via the following measures:
  A. Distal vertical situation of the bone plateau compared to the implant by retroalveolar radiography
  B. Mesial vertical situation of the bone plateau compared to the implant by retroalveolar radiography
  C. Insertion Torque Value (Ncm)
  These changes are evaluated from Baseline to Visit 3.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Hoornaert, DDS, Principal Investigator — University Hospital of Nantes
Locations (9):
- France (9):
  - Hospital University of Nantes, Nantes
  - Private dental practice office of Dr. Alain Hoornaert, Nantes
  - Private dental practice office of Dr. Samer Saloum-Rouxel, Nantes
  - Private dental practice office of Dr. Xavier Struillou, Nantes
  - Private dental practice office of Dr. Edouard Lanoiselée, Nozay
  - Private dental practice office of Dr. Aurélien Fruchet, Olonne-sur-Mer
  - Private dental practice office of Dr. Hélène Le Hécho, Orée d'Anjou
  - Private dental practice office of Dr. Nicolas Strube, Orvault
  - Private dental practice office of Dr. Romain Besnier, Orvault

IPD SHARING:
Plan to Share IPD: No